CLINICAL TRIAL: NCT02115425
Title: Samsung Bioimpedance System Calibration Study
Brief Title: Calibrate Samsung's BIA to Meseaure Body Composition
Acronym: Samsung
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Samsung (Industry)
Responsible Party: Principal Investigator, Jolene Zheng, Principal investigator, Pennington Biomedical Research Center
Other Study IDs: PBRC 2014-005
Record Dates: First submitted 2014-04-14; First posted 2014-04-16 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Body Composition; Circumference Measurements; Tissue Thickness Measurements
MeSH Terms: interventions — Body Weights and Measures; Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Age 10-17: Participants age 5 - 17 will complete the following Body Measurements Body Composition and Circumference Measurements Whole Body DXA Scan Bioelectrical Impedance Analysis (BIA)
  Interventions: Other: Body Measurements; Other: Whole Body DXA Scan; Other: Bioelectrical Impedance Analysis (BIA); Other: add name here
- Age 18-80: Age 18-80 years Participants age 18-80 will complete the following Body Measurements Body Composition and Circumference Measurements Whole Body DXA Scan Bioelectrical Impedance Analysis (BIA)
  Interventions: Other: Body Measurements; Other: Whole Body DXA Scan; Other: Bioelectrical Impedance Analysis (BIA); Other: add name here

INTERVENTIONS:
Other: Body Measurements — A series of body measurements will be taken by trained staff. These measurements include height and weight. These measurements will be completed twice during this time. You will wear a hospital gown and bathing suit for these measurements.
Other: Whole Body DXA Scan — This scan measures the amount of bone, muscle, and fat in your body. The scan will be performed using a whole-body scanner. You will be required to wear a hospital gown, to remove all metal-containing objects from your body, and to lie down on the table.
  Other Names: Dual-energy X-ray Absorptiometry Scan
Other: Bioelectrical Impedance Analysis (BIA) — These tests will measure the amount of fat in your body. You will be asked to change into a hospital gown and to remove all footwear and socks/stockings. Once changed and barefoot, you will be asked to stand on a scale (similar to a large gym scale) and to hold on to hand electrodes on each side of the scale. You will be asked to step off of the scale once the measurement is complete (less than one minute). You will also hold on to hand electrodes for three other BIA systems.
  Other Names: InBody720; http://www.biospaceamerica.com/Product/ib720.html
Other: Bioelectrical Impedance Analysis (BIA) — These tests will measure the amount of fat in your body. You will be asked to change into a hospital gown and to remove all footwear and socks/stockings. You will be asked to hold on to hand electrodes on a hand hold device. You will be asked to complete 3 measurement (less than one minute). You will also hold on to hand electrodes for two other BIA systems.
  Other Names: Omron 214; Omron 510; Omron 306
Other: add name here

SUMMARY:
The purpose of this study is to collect body composition data using bioimpedance analysis (Samsung) and DXA (GE Medical). Both of the methods are explained in more detail in section 5 of this consent. The data collected will help Samsung improve the products the company offers.

DETAILED DESCRIPTION:
If you are eligible and you choose to participate in this study, you will be asked to come to the Bone & Joint Clinic of Baton Rouge in Baton Rouge between 7:00 and 11:00 am after at least a two-hour fast (nothing to eat or drink besides water for 2 hours prior to your appointment). You will be asked not to exercise, shower, or use a steam room or sauna at least two hours prior to evaluation. The study visit will take approximately one hour. During the visit, you will complete the informed consent process and then complete the baseline body measurements and body composition procedures immediately afterwards. Adult pre-menopausal women will have a urine pregnancy test prior to evaluation. Study procedures are not for diagnostic or treatment purposes and the DXA scan is intended for research purposes.

Description of study procedures

Body Measurements (about 15 minutes):

A series of body measurements will be taken by trained staff. These measurements include height, weight, and vital signs. The weight and height measurements will be completed twice during this time. The subject will wear a hospital gown and tight fitting garments for these procedures and the subject's BMI will be calculated from these measurements.

Body Composition Measurements

Whole Body DXA Scan, about 20 minutes This scan measures the amount of bone, muscle, and fat in your body. The scan will be performed using a whole-body scanner. The subject will be required to wear a hospital gown, to remove all metal-containing objects from the body, and to lie down on the table. The subject will be carefully positioned on the table, and the legs will be placed together using two Velcro straps. A scanner emitting low energy X-rays and a detector will pass along the body. The subject will be asked to remain completely still while the scan is in progress. The scan takes approximately ten minutes.

Impedance Analysis (BIA) (about 10 minutes):

These tests will measure the amount of fat in the body. These procedures will vary depending on the measurement system and several different BIA systems will be used during this test.

Some examples are presented in the supplementary material at the end of this protocol.

Specifically, the following systems will be used in this study:

Samsung Health Cover; Measure 3 times; Standing Posture

Marketed systems:

InBody720 (http://www.biospaceamerica.com/Product/ib720.html; measure one time; Standing Posture Omron 306; Measure 1 time; Standing Posture Omron 510; Measure 1 time; Standing Posture

ELIGIBILITY:
Inclusion Criteria:

* Being either male or female
* Being from 18 to 80 years of age
* Being considered underweight, normal weight, overweight, or obese based on specified BMI ranges
* Having a body weight of less than 440 pounds
* Being willing to comply with the study procedures
* Females must not be pregnant, breastfeeding, or planning to become pregnant within the next 6 months.

Exclusion Criteria:

* Being Asian. Note that Asian subjects have already been evaluated as part of the Korean phase of this investigation.
* Having a significant chronic disease as judged by the investigator
* Having metal-containing objects in your body
* Being pregnant or attempting to become pregnant
* Having medical implants such as a pacemaker or metal joint replacements
* Being a professional athlete or someone with severe edema or dehydration
* Having a body weight greater than 440 pounds
* Being a body builder as judged by the investigator
* Adults unable to consent
* Prisoners

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Male or Female age 10-80 years of age.
Sampling Method: Probability Sample
Enrollment: 421 (Actual)
Dates: Start 2014-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Calibrate the Samsung BIA System by collecting body composition using two different methods and 5 different equipment | First Visit (Only one visit)
  The study will be conducted in two overlapping phases. In Phase I, approximately 300 adult subjects (>18 to 80 yrs, equal numbers of female and male) will be recruited to take part in this study as detailed below: (1) Underweight (BMI<18.5 k/m2), 50 subjects. (2) Normal-Overweight (18.5-30), 150 subjects. (3) Obese (>30), 100 subjects.
  Phase II, planned to start later this spring and summer, will involve evaluation of children and 100 subjects (10-</=18 yrs, equal numbers of female and male) are planned in this phase as: (1) Normal-Overweight (18.5-30), 50 subjects. (2) Obese (>30), 50 subjects. An addendum describing details of this study phase will be forthcoming.
  Informed consent for both adults and children will be obtained for this study. Written and verbal assents for children will be obtained for this study.

SECONDARY OUTCOMES:
Improve the BIA body composition predictions using circumference and tissue thickness measurements | First Visit (Only one visit)
  Part II: Verify developed algorithms:
  * Task A: Body Fat Analysis
  * Task B: Body Muscle Analysis
  * Task C: TBW (total body water), ICW (intracellular water), ECW (extracelluar water)

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States